CLINICAL TRIAL: NCT06768762
Title: Optimizing a Remote-based Physical Activity Intervention for Adults with Total Knee Replacement
Acronym: MOST Energized
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christine A Pellegrini, PhD, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00136251; R01AG088083 (NIH)
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Knee Replacement
Keywords: knee replacement; exercise; online
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- Experimental condition 1 (Experimental): Energize Online Program plus phone coaching, progress reports to physicians, 'Hear From Others' videos, and individualized feedback
  Interventions: Behavioral: Phone Coaching; Behavioral: Progress reports to providers; Behavioral: 'Hear from Others' Videos; Behavioral: Individualized Feedback; Behavioral: Online exercise program
- Experimental condition 2 (Experimental): Energize Online Program plus phone coaching, progress reports to physicians, and 'Hear From Others' videos
  Interventions: Behavioral: Phone Coaching; Behavioral: Progress reports to providers; Behavioral: 'Hear from Others' Videos; Behavioral: Online exercise program
- Experimental condition 3 (Experimental): Energize Online Program plus phone coaching, progress reports to physicians, and individualized feedback
  Interventions: Behavioral: Phone Coaching; Behavioral: Progress reports to providers; Behavioral: Individualized Feedback; Behavioral: Online exercise program
- Experimental condition 4 (Experimental): Energize Online Program plus phone coaching and progress reports to physicians
  Interventions: Behavioral: Phone Coaching; Behavioral: Progress reports to providers; Behavioral: Online exercise program
- Experimental condition 5 (Experimental): Energize Online Program plus phone coaching, 'Hear From Others' videos, and individualized feedback
  Interventions: Behavioral: Phone Coaching; Behavioral: 'Hear from Others' Videos; Behavioral: Individualized Feedback; Behavioral: Online exercise program
- Experimental condition 6 (Experimental): Energize Online Program plus phone coaching and 'Hear From Others' videos
  Interventions: Behavioral: Phone Coaching; Behavioral: 'Hear from Others' Videos; Behavioral: Online exercise program
- Experimental condition 7 (Experimental): Energize Online Program plus phone coaching and individualized feedback
  Interventions: Behavioral: Phone Coaching; Behavioral: Individualized Feedback; Behavioral: Online exercise program
- Experimental condition 8 (Experimental): Energize Online Program plus phone coaching
  Interventions: Behavioral: Phone Coaching; Behavioral: Online exercise program
- Experimental condition 9 (Experimental): Energize Online Program plus progress reports to physicians, 'Hear From Others' videos, and individualized feedback
  Interventions: Behavioral: Progress reports to providers; Behavioral: 'Hear from Others' Videos; Behavioral: Individualized Feedback; Behavioral: Online exercise program
- Experimental condition 10 (Experimental): Energize Online Program plus progress reports to physicians and 'Hear From Others' videos
  Interventions: Behavioral: Progress reports to providers; Behavioral: 'Hear from Others' Videos; Behavioral: Online exercise program
- Experimental condition 11 (Experimental): Energize Online Program plus progress reports to physicians and individualized feedback
  Interventions: Behavioral: Progress reports to providers; Behavioral: Individualized Feedback; Behavioral: Online exercise program
- Experimental condition 12 (Experimental): Energize Online Program plus progress reports to physicians
  Interventions: Behavioral: Progress reports to providers; Behavioral: Online exercise program
- Experimental condition 13 (Experimental): Energize Online Program plus 'Hear From Others' videos and individualized feedback
  Interventions: Behavioral: 'Hear from Others' Videos; Behavioral: Individualized Feedback; Behavioral: Online exercise program
- Experimental condition 14 (Experimental): Energize Online Program plus 'Hear From Others' videos
  Interventions: Behavioral: 'Hear from Others' Videos; Behavioral: Online exercise program
- Experimental condition 15 (Experimental): Energize Online Program plus individualized feedback
  Interventions: Behavioral: Individualized Feedback; Behavioral: Online exercise program
- Experimental condition 16 (Experimental): Energize Online Program
  Interventions: Behavioral: Online exercise program

INTERVENTIONS:
Behavioral: Phone Coaching — Participants will receive 11 coaching calls with a health coach. Calls will occur weekly during the first month, twice/month during months 2-3, and once/month during months 4-6. Each call is expected to last 10-15 minutes.
  Arms: Experimental condition 1; Experimental condition 2; Experimental condition 3; Experimental condition 4; Experimental condition 5; Experimental condition 6; Experimental condition 7; Experimental condition 8
Behavioral: Progress reports to providers — Progress reports on physical activity and program adherence will be sent to participants providers at 3 and 6 months.
  Arms: Experimental condition 1; Experimental condition 10; Experimental condition 11; Experimental condition 12; Experimental condition 2; Experimental condition 3; Experimental condition 4; Experimental condition 9
Behavioral: 'Hear from Others' Videos — Participants will receive monthly 'Hear From Others' videos. The videos will include other adults with knee replacement discussing the challenges they have faced and strategies to overcome barriers to activity.
  Arms: Experimental condition 1; Experimental condition 10; Experimental condition 13; Experimental condition 14; Experimental condition 2; Experimental condition 5; Experimental condition 6; Experimental condition 9
Behavioral: Individualized Feedback — Participants will receive individualized feedback from a coach via email. The feedback will specifically focus on participant responses to the 'Apply Your Knowledge' activities and will correspond with the video lessons. Feedback will be weekly during months 1-3 and monthly during months 4-6.
  Arms: Experimental condition 1; Experimental condition 11; Experimental condition 13; Experimental condition 15; Experimental condition 3; Experimental condition 5; Experimental condition 7; Experimental condition 9
Behavioral: Online exercise program — MOST Energized! Online Exercise Program

SUMMARY:
The purpose of this study is to identify which supplemental intervention components added to an online exercise program contribute to the greatest increases in physical activity (total MVPA and percent meeting guidelines [≥150 min/week of MVPA]) in adults with knee replacement at 6 and 12 months. Secondary outcomes will examine changes in pain and physical function.

DETAILED DESCRIPTION:
All participants will receive a 6-month, fully automated online behavioral exercise program (Energize! Exercise Program). This program is designed to increase moderate-intensity physical activity among individuals who engage in little to no physical activity at baseline. Over the course of the program, participants are given a physical activity goal which starts at 75 minutes per week and gradually progresses to 200 minutes per week. Participants are instructed to view a 10-15-minute video lesson weekly, during months 1-3, and monthly during months 4-6. These lessons teach behavioral principles for increasing exercise and maintaining physical activity long-term. Participants are also asked to complete an 'Apply Your Knowledge' activity after watching each video lesson. These activities are designed to help the participant engage more with the lesson content, with a particular emphasis on applying the content to their lives. Within this program, participants are also asked to plan and report their exercise each week, and automated feedback is provided based upon their weekly physical activity reports.

In addition to receiving the Energize! Exercise Program, participants will be randomly assigned to receive 0-4 supplemental intervention components (phone coaching, progress reports to providers, 'Hear From Others' videos, and individualized feedback) which are each described in more detail below.

ELIGIBILITY:
Inclusion Criteria:

* had a knee replacement (including primary, staged or independent bilateral, or revision) at least 12 months ago
* have a computer, tablet, or smartphone with active internet access
* self-report engaging in less than 60 minutes/week of moderate-intensity physical activity
* be English-speaking and able to read consent and study materials written in English
* be willing to complete the 4 remote assessments, including physical activity monitoring
* be willing to be randomized to receive 0-4 supplemental intervention components.

Exclusion Criteria:

* any contraindications to physical activity (e.g., chest pain)
* have a scheduled surgery within the next 12 months (e.g., hip or knee replacement)
* have a mobility limiting comorbidity unrelated to knee replacement
* live outside of the continental U.S
* do not currently have a physician or orthopedic surgeon whom they see regularly
* are currently participating in physical therapy (for knee)
* are participating in a structured weight loss or physical activity program
* unable to provide proof of knee replacement surgery
* have a BMI >40kg/m2
* score >30 on PROMIS cognitive function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity (min/week) | Baseline to 6 months
  Change in Actigraph-assessed moderate-to-vigorous intensity physical activity
Percentage meeting physical activity guidelines | 6 months
  Percentage of participants meeting physical activity guidelines (150 minutes/week)
Physical activity (min/week) | Baseline to 12 months
  Change in Actigraph-assessed moderate-to-vigorous intensity physical activity
Percentage meeting physical activity guidelines | 12 months
  Percentage of participants meeting physical activity guidelines (150 minutes/week)

SECONDARY OUTCOMES:
Pain intensity | Baseline to 6 months
  Change in pain intensity using Patient-Reported Outcomes Measurement Information System (PROMIS)
Physical Function | Baseline to 6 months
  Change in physical function using the physical function/mobility Patient-Reported Outcomes Measurement Information System (PROMIS)
Pain intensity | Baseline to 12 months
  Change in pain intensity using Patient-Reported Outcomes Measurement Information System (PROMIS)
Physical Function | Baseline to 12 months
  Change in physical function using the physical function/mobility Patient-Reported Outcomes Measurement Information System (PROMIS)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Pellegrini, PhD, Principal Investigator — University of South Carolina; Jessica Unick, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be deposited into Zenodo at either the time of associated publication or the end of the performance period
Supporting Information: Study Protocol, SAP, ICF